CLINICAL TRIAL: NCT04748627
Title: Global IBD Visualization of Epidemiology Studies (GIVES) in the 21st Century (GIVES-21)
Brief Title: Global IBD Visualization of Epidemiology Studies (GIVES) in the 21st Century
Acronym: GIVES-21
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: GIVES-21
Record Dates: First submitted 2021-02-09; First posted 2021-02-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Crohn's disease (CD) and Ulcerative colitis (UC) are chronic inflammatory bowel diseases (IBD) of unknown etiology. The pathophysiology of IBD relates to the mucosal immune response to antigenic stimulation from the gut microbiota secondary to environmental influence, on a background of genetic susceptibility. IBD represents an important public health problem because it affects mostly young people at an age when they are most active in their private and professional life, and a management challenge because of its unpredictable relapsing nature. During the last few decades the incidence of IBD has changed in many ways. Incidence rates of traditionally high incidence areas such as the United States and Europe is remaining relatively stable or even decreasing, while the diseases have become more prevalent in previously low incidence areas, including Asia. Our latest systematic review has demonstrated that the highest reported prevalence of IBD was still in Europe and North America, however, the incidence of IBD has been rising in newly industrialized countries since 1990.

DETAILED DESCRIPTION:
Investigators aim to study the incidence, demographic factors, and disease outcomes of IBD patients, environmental and dietary factors associated with IBD in 19 regions globally. Via the web registration, investigators intend to form a new prospective, uniformly diagnosed, population-based inception cohort of patients with IBD. Physicians, gastroenterologists, family doctors, surgeons and pathologists in the study area will be notified repeatedly about the study by letter, telephone, internet, personal visit of the investigators, and encouraged to inform investigators of every possible new case of IBD. Endoscopic, pathology and radiology records will be canvassed repeatedly for likely cases, both electronically and manually. By these methods, investigators intend to capture over 90% of possible cases. All patients are required to meet the diagnostic criteria for IBD on the basis of clinical symptoms, endoscopic or radiological evidence or mucosal biopsies. Infectious gastroenteritis, tuberculosis, entamoeba and cancer have to be ruled out. The web-based database application will be used for online registration of the various registration forms and questionnaires and the database is located on a central secured server. With the data collected, an online interactive atlas will be created which allows the community to visualize the most up-to-date epidemiology of IBD with the aims to promotes knowledge translation and research endeavours of stakeholders and provide infrastructure, resources, and expertise to define Crohn's disease burden in regions of the world where the disease is emerging.

ELIGIBILITY:
For IBD patients:

Inclusion Criteria:

* Aged ≥ 18 years old
* Confirmed diagnosis of Crohn's disease or Ulcerative Colitis according to established clinical, endoscopic and histological criteria
* Written informed consent obtained

Exclusion Criteria:

* Nil

For healthy control:

Inclusion criteria:

* Aged ≥ 18 years old
* Asymptomatic
* Written informed consent obtained

Exclusion Criteria:

* Diagnosis of any chronic medical illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For IBD patients:
  Newly diagnosed IBD patients in the local area
  For heathy control:
  Asymptomatic adults who have no IBD or any other chronic medical illnesses.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of IBD | 1 year
  To determine the incidence of IBD in 19 regions globally, and to investigate if this increase is caused by environmental and dietary factors.

SECONDARY OUTCOMES:
Geographical effect | 1 year
  To study the geographical effect on: 5-amino-salicylic acid, corticosteroids, immunosuppressive agents, biologics and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong